CLINICAL TRIAL: NCT00356031
Title: A Phase II Study of Neoadjuvant Bevacizumab and Radiation Therapy for Resectable Soft Tissue Sarcomas
Brief Title: Bevacizumab and Radiation Therapy for Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yen-Lin Evelyn Chen, MD, Study Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-090; 1R21CA117128-01A1 (NIH)
Record Dates: First submitted 2006-07-21; First posted 2006-07-25 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Soft Tissue Sarcoma; Fibrous Histiocytoma; Liposarcoma; Leiomyosarcoma; Fibrosarcoma; Synovial Sarcoma
Keywords: Avastin
MeSH Terms: conditions — Sarcoma; Histiocytoma, Benign Fibrous; Liposarcoma; Leiomyosarcoma; Fibrosarcoma; Sarcoma, Synovial | interventions — Bevacizumab; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab, Radiation, and Surgery (Experimental): Bevacizumab 5mg/kg, external beam radiation therapy (XRT), surgery, Intraoperative radiation therapy (IORT), and postoperative external beam radiation therapy (Post-op XRT)
  Interventions: Drug: Bevacizumab; Radiation: Radiation Therapy; Procedure: Surgery

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 5mg/kg given intravenously every 2 weeks for a total of 4 doses
  Other Names: Avastin
Radiation: Radiation Therapy — External beam radiation given two weeks after the first bevacizumab infusion and delivered 5 days a week at 1.8 Gy per day, over 6 weeks. Total radiation dose is 50.4 Gy. For patients with tumors in the retroperitoneum or pelvis, intraoperative radiation therapy (10-20 Gy) may be given for close or positive margins at the discretion of the radiation oncologist and surgeon. For patients with tumors in the extremity or trunk, post-operative external beam radiation therapy (10-20 Gy) will be given for close or positive margins assuming wound healing is good.
Procedure: Surgery — Surgical resection is performed 6-7 weeks after completion of neoadjuvant therapy.

SUMMARY:
The main purpose of this study is to test the effectiveness of bevacizumab in combination with radiation therapy to see what effects (good or bad) they have on patients with soft tissue sarcoma. Bevacizumab is an antibody designed specifically to slow or stop the growth of cancerous tumors by decreasing the blood supply to the tumor. Bevacizumab is approved by the FDA in combination with intravenous 5-fluorouracil-based chemotherapy as a treatment for patients with cancer of the colon or rectum that has spread. However, the use of bevacizumab in combination with radiation for sarcomas is still under investigation.

DETAILED DESCRIPTION:
* The dose of bevacizumab and radiation therapy will be the same for all participants throughout the study.
* Bevacizumab will be given as an intravenous infusion every 2 weeks for a total of 4 doses.
* Radiation therapy will begin 2 weeks after the first bevacizumab infusion and will be delivered 5 days per week over a period of 6 weeks. This is done as an outpatient procedure. Each 2 week period will be considered a separate treatment cycle. Participants will be treated with radiation therapy for a maximum of 3 cycles (6 weeks).
* A surgeon will evaluate the participants tumor by radiologic studies before study treatment to determine if surgical removal is possible. After the completion of study treatment, a surgeon will repeat the evaluation of the tumor. Surgery will performed 6-7 weeks after the completion of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary soft tissue sarcoma (STS) or an isolated local recurrence of STS. Open incisional biopsy or core biopsies should be performed within 8 weeks prior to registration
* Tumor grade of intermediate or high grade
* Tumor must be located on the upper extremity, the lower extremity, trunk, retroperitoneum, or pelvis
* Primary tumors must be > 5.0cm in maximal diameter and local recurrence can be any size
* 18 years of age or older
* Zubrod performance status of 0-2
* Adequate organ and marrow function

Exclusion Criteria:

* Metastatic disease
* Pregnant or lactating women
* HIV positive patients
* Prior treatment with radiation, chemotherapy or biotherapy for this tumor
* History or evidence of central nervous system (CNS) disease
* Serious, non-healing wound, ulcer, or bone fracture
* Clinically significant cardiovascular disease, New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or Grade II or greater peripheral vascular disease within 1 year
* History of stroke within the past 6 months
* Major surgical procedure or significant traumatic injury within 28 days
* Current or recent (within 10 days) use of full-dose oral or parenteral anticoagulants or thrombolytic agents.
* Presence of bleeding diathesis or coagulopathy
* Proteinuria at baseline or clinically significant impairment of renal function
* History of abdominal fistula, gastrointestinal perforation, or inta-abdominal abscess within the past 6 months
* Documented history of uncontrolled seizures
* Grade 2 or greater sensory neuropathy based upon the NCI CTCAE, version 3.0
* Known history of deep vein thrombosis or pulmonary embolus
* Known hypercoagulable disorder
* History of hepatic cirrhosis or current hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Lin Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Yoon SS, Duda DG, Karl DL, Kim TM, Kambadakone AR, Chen YL, Rothrock C, Rosenberg AE, Nielsen GP, Kirsch DG, Choy E, Harmon DC, Hornicek FJ, Dreyfuss J, Ancukiewicz M, Sahani DV, Park PJ, Jain RK, Delaney TF. Phase II study of neoadjuvant bevacizumab and radiotherapy for resectable soft tissue sarcomas. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):1081-90. doi: 10.1016/j.ijrobp.2010.07.024. Epub 2010 Oct 6. PMID 20932656
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the multidisciplinary sarcoma clinic, surgical oncology, radiation oncology, and medical oncology clinics at the Massachusetts General Hospital, Brigham and Women's Hospital, or Dana-Farber Cancer Institute.
Groups:
- Experimental: Bevacizumab, Radiation, and Surgery: Bevacizumab 5mg/kg, external beam radiation therapy (XRT), surgery, Intraoperative radiation therapy (IORT), and postoperative external beam radiation therapy (Post-op XRT)
  Bevacizumab: Bevacizumab 5mg/kg given intravenously every 2 weeks for a total of 4 doses
  Radiation Therapy: External beam radiation given two weeks after the first bevacizumab infusion and delivered 5 days a week at 1.8 Gy per day, over 6 weeks. Total radiation dose is 50.4 Gy. For patients with tumors in the retroperitoneum or pelvis, intraoperative radiation therapy (10-20 Gy) may be given for close or positive margins at the discretion of the radiation oncologist and surgeon. For patients with tumors in the extremity or trunk, post-operative external beam radiation therapy (10-20 Gy) will be given for close or positive margins assuming wound healing is good.
  Surgery: Surgery is performed 6-7 weeks after completion of neoadjuvant therapy.
Period: Overall Study
Arm/Group | Experimental: Bevacizumab, Radiation, and Surgery
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bevacizumab, Radiation, and Surgery: Bevacizumab 5mg/kg, external beam radiation therapy (XRT), surgery, Intraoperative radiation therapy (IORT), and postoperative external beam radiation therapy (Post-op XRT)
  Bevacizumab: Bevacizumab 5mg/kg given intravenously every 2 weeks for a total of 4 doses
  Radiation Therapy: External beam radiation given two weeks after the first bevacizumab infusion and delivered 5 days a week at 1.8 Gy per day, over 6 weeks. Total radiation dose is 50.4 Gy. For patients with tumors in the retroperitoneum or pelvis, intraoperative radiation therapy (10-20 Gy) may be given for close or positive margins at the discretion of the radiation oncologist and surgeon. For patients with tumors in the extremity or trunk, post-operative external beam radiation therapy (10-20 Gy) will be given for close or positive margins assuming wound healing is good.
  Surgery: Surgery is performed 6-7 weeks after completion of neoadjuvant therapy.
Arm/Group | Bevacizumab, Radiation, and Surgery
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 20
Sarcoma Histology [Count of Participants; unit: Participants]
  Fibroblastic | 8
  Liposarcoma | 6
  Leiomyosarcoma | 4
  Fibroblastic Osteosarcoma | 1
  Not Otherwise Specified | 1
Sarcoma Grade [Count of Participants; unit: Participants]
  Low | 2
  Intermediate | 8
  High | 10
Median Sarcoma Size [Median (Full Range); unit: Centimeters (cm)] | 8.25 [5 to 20.2]
Sarcoma Location [Count of Participants; unit: Participants]
  Extremity | 13
  Trunk | 1
  retroperitoneal/pelvis tumors | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate for Neoadjuvant Bevacizumab Combined With Radiation Therapy for Intermediate and High-risk Soft Tissue Sarcomas.
Description: The count of participants with greater than or equal to 80% pathological necrosis in the resected specimen following neoadjuvant bevacizumab and radiation.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Bevacizumab, Radiation, and Surgery
Number analyzed (Participants) | 20
participants
  80-89% necrosis | 2
  90-99% necrosis | 4
  100% necrosis | 3

2. Secondary Outcome: Change in Median Microvessel Density (MVD) After Bevacizumab Alone
Description: The percentage change in median microvessel density (MVD) after Bevacizumab treatment alone
Time Frame: baseline and 3 years
Measure: Median (95% Confidence Interval); unit: percentage of change in MVD
Arm/Group | Bevacizumab, Radiation, and Surgery
Number analyzed (Participants) | 20
percentage of change in MVD | 53 [28.6 to 77.4]
Statistical Analysis 1: Comparison: Bevacizumab, Radiation, and Surgery; Test type: Other; p < .05, t-test, 1 sided

3. Secondary Outcome: Average Change in Blood Flow, Blood Volume,and Permeability Surface Area
Description: The percentage reduction in blood flow, blood volume,and permeability surface area of the tumor following combination therapy as determined by perfusion CT (computerized tomography) scan. The percent change represents the combined average percent change for flow, volume, and permeability together.
Time Frame: 3 years
Measure: Mean (Full Range); unit: Percent Reduction
Arm/Group | Bevacizumab, Radiation, and Surgery
Number analyzed (Participants) | 20
Percent Reduction | 67 [62 to 72]
Statistical Analysis 1: Comparison: Bevacizumab, Radiation, and Surgery; Test type: Other; p < .05, t-test, 1 sided

4. Secondary Outcome: Local Control Rate
Description: The number of patients with local recurrence after a median follow-up of 24 months. Local recurrence is defined as disease progression (new cancer growth) at the primary cancer site.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab, Radiation, and Surgery
Number analyzed (Participants) | 20
Participants
  Local Recurrence | 1
  No Local Recurrence | 19

5. Secondary Outcome: Distant Recurrence
Description: The number of participants with distant recurrence at the time of last follow-up. Distant recurrence is when cancer has spread (metastasized) to areas farther away from where the primary cancer site is.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Bevacizumab, Radiation, and Surgery
Number analyzed (Participants) | 20
Participants
  Distant recurrence | 7
  No distant recurrence | 13

6. Secondary Outcome: Disease Free Survival
Description: The median amount of time from the end of treatment until to distant recurrence. Distant recurrence is when cancer spreads to areas in the body away from the primary cancer site.
Time Frame: 3 years
Measure: Median (Full Range); unit: Months
Arm/Group | Experimental: Bevacizumab, Radiation, and Surgery
Number analyzed (Participants) | 20
Months | 7 [2 to 36]

ADVERSE EVENTS:
Time Frame: 3 years
Description: Laboratory tests and physical exams were performed as a part of routine study visits.
Arm/Group | Bevacizumab, Radiation, and Surgery
All-Cause Mortality (participants affected / at risk) | 3/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab, Radiation, and Surgery (N=20)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Dyspnea (Reproductive system and breast disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab, Radiation, and Surgery (N=20)
Allergic reaction (Immune system disorders) | 3 (12)
Allergic rhinitis (Immune system disorders) | 3 (5)
Hemoglobin (Blood and lymphatic system disorders) | 10 (23)
Leukocytes (Blood and lymphatic system disorders) | 3 (15)
Lymphopenia (Blood and lymphatic system disorders) | 7 (21)
Neutrophils (Blood and lymphatic system disorders) | 3 (5)
Platelets (Blood and lymphatic system disorders) | 2 (4)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 10 (49)
Hypotension (Cardiac disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 11 (40)
Fever w/o neutropenia (General disorders) | 2 (2)
Insomnia (General disorders) | 4 (5)
Partial thromboplastin time (Blood and lymphatic system disorders) | 3 (4)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (9)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 3 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (5)
Wound - non-infectious (Skin and subcutaneous tissue disorders) | 2 (2)
Skin-other (Skin and subcutaneous tissue disorders) | 5 (17)
Anorexia (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (5)
Dehydration (Gastrointestinal disorders) | 1 (2)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 6 (10)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1 (4)
Nausea (Gastrointestinal disorders) | 8 (12)
Taste disturbance (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
GI-other (Gastrointestinal disorders) | 2 (4)
Hematoma (Blood and lymphatic system disorders) | 2 (2)
Nose, hemorrhage (Blood and lymphatic system disorders) | 3 (6)
Hemorrhage-other (Blood and lymphatic system disorders) | 1 (1)
Infection Gr0-2 neut, skin (Infections and infestations) | 1 (2)
Infection Gr0-2 neut, stomach (Infections and infestations) | 1 (1)
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1 (1)
Infection Gr0-2 neut, vagina (Infections and infestations) | 1 (1)
Infection Gr0-2 neut, wound (Infections and infestations) | 1 (2)
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 1 (2)
Edema limb (Blood and lymphatic system disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (18)
ALT, SGPT (Metabolism and nutrition disorders) | 2 (8)
AST, SGOT (Metabolism and nutrition disorders) | 3 (8)
Bilirubin (Metabolism and nutrition disorders) | 1 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (28)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Proteinuria (Metabolism and nutrition disorders) | 4 (12)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5)
Metabolic/Laboratory-other (Metabolism and nutrition disorders) | 1 (12)
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue necrosis, extremity lower (Musculoskeletal and connective tissue disorders) | 1 (3)
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 3 (8)
Anxiety (Nervous system disorders) | 1 (4)
Depression (Nervous system disorders) | 3 (5)
Neuropathy-sensory (Nervous system disorders) | 2 (11)
Neurologic-other (Nervous system disorders) | 1 (2)
Abdomen, pain (General disorders) | 1 (1)
Back, pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Chest/thoracic pain NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 3 (8)
Head/headache (General disorders) | 3 (7)
Joint, pain (Musculoskeletal and connective tissue disorders) | 3 (8)
Pelvic, pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Skin, pain (Skin and subcutaneous tissue disorders) | 1 (1)
Throat/pharynx/larynx, pain (Gastrointestinal disorders) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pain-other (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Irregular menses (Reproductive system and breast disorders) | 2 (4)
Tumor lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Visceral arterial ischemia (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of patients. Results require validation in a larger cohort of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No